CLINICAL TRIAL: NCT03995602
Title: A Randomised, Placebo-controlled, Crossover Study of the Effects of Dragon Fruit Effects of Dragon Fruit (Pitaya) Consumption on Vascular Function in Healthy Males and Females
Brief Title: The Effects of Dragon Fruit Consumption on Vascular Function.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Dr Ana Rodriguez-Mateos, Lecturer in Nutritional Sciences, King's College London
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: DRAGON Study
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Healthy Men and Women
Keywords: vascular function; endothelial function; betalains; dragon fruit; pitaya

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dragon fruit first then placebo (Experimental): 2 weeks of dragon fruit juice intake or placebo with crossover to the other
  Interventions: Dietary Supplement: Dragon fruit juice drink; Dietary Supplement: Placebo
- Placebo first then dragon fruit (Experimental): 2 weeks of dragon fruit juice intake or placebo with crossover to the other
  Interventions: Dietary Supplement: Dragon fruit juice drink; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Dragon fruit juice drink — Dragon fruit drink containing 24 g of freeze-dried dragon fruit powder dissolved in low nitrate water.
Dietary Supplement: Placebo — Drink with macro- and micro-nutrient matched against the intervention drink.

SUMMARY:
Native to South America and South East Asia, the dragon fruit (pitaya) has become increasingly popular world-wide due to their vivid hue and bizarre structure. More importantly, their high levels of bioactive phytochemical betalains has sparked considerable scientific interest. Recent findings from in vitro and in vivo animal studies tentatively suggest that betalains may have ameliorative effects on vascular function. This will be a first randomised controlled trial aimed to explore the impact of dragon fruit consumption on blood pressure and other vascular parameters in healthy individuals. The study will feature a randomised, double-blinded, placebo-controlled and crossover design with flow-mediated dilatation (FMD) as primary outcome along with blood pressure and arterial stiffness as secondary outcomes. Cardiovascular biomarkers as well as relevant metabolites will also be determined from blood and urine samples collected from participants.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women aged 18-40 years old
2. Subjects are willing to maintain their normal eating/drinking habits and exercise habits to avoid changes in body.

   weight over the duration of the study.
3. Are able to understand the nature of the study.
4. Able to give signed written informed consent.
5. Signed informed consent form.

Exclusion Criteria:

1. Medical history of cardiovascular disease including coronary artery disease, cerebrovascular disease and peripheral artery disease.
2. Hypertensive, as defined as SBP superior or equal to 140 mmHg.
3. Obese participants, defined as BMI superior or equal to 30.
4. Medical history of diabetes mellitus, metabolic syndrome, terminal renal failure or malignancies.
5. Abnormal heart rhythm (lower or higher than 60-100 bpm).
6. Allergies to dragon fruit, cactus pear or other significant food allergy.
7. Subjects under medication that can affect the cardiovascular system or on vitamin/dietary supplements.
8. Subjects who have lost more than 10% of their weight in the past 6 months or are currently in a diet
9. Subjects who reported participant in another study within one month before the study start.
10. Subjects who smokes.
11. Pregnant women or planning to become pregnant in the next 6 months.
12. Any reason or condition that in the judgment of the clinical investigator(s) may put the subject at unacceptable risk or that may preclude the subject from understanding or complying with the study's requirements.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Changes in flow mediated dilation (FMD) of the brachial artery | Baseline & 2 weeks
  Determine changes in flow mediated dilation (FMD) of the brachial artery after 2 weeks consumption of 24 g freeze-dried dragon fruit.

SECONDARY OUTCOMES:
Changes in flow mediated dilation (FMD) of the brachial artery | Baseline & 2, 3 and 4 hour post-consumption
  Determine changes in flow mediated dilation (FMD) of the brachial artery at 2, 3, and 4 hour post consumption of 24 g freeze-dried dragon fruit.
Changes in blood pressure | Baseline & 2, 3 and 4 hour post-consumption
  Determine changes in systolic and diastolic blood pressure at 2, 3, and 4 hour post consumption of 24 g freeze-dried dragon fruit.
Changes in blood pressure | Baseline & 2 weeks
  Determine changes in systolic and diastolic blood pressure after 2 weeks post consumption of 24 g freeze-dried dragon fruit.
Changes in heart rate | Baseline & 2, 3 and 4 hour and 2 weeks post-consumption
  Determine changes in heart rate post consumption of 24 g freeze-dried dragon fruit.
Changes blood flow velocity | Baseline & 2, 3 and 4 hour and 2 weeks post-consumption
  Determine changes in blood flow velocity post consumption of 24 g freeze-dried dragon fruit.
Changes in pulse wave velocity (PWV) | Baseline & 3 hour and 2 weeks post-consumption.
  Determine changes in pulse wave velocity post consumption of 24 g freeze-dried dragon fruit.
Changes augmentation Index (AIx) | Baseline & 3 hour and 2 weeks post-consumption.
  Determine changes in augmentation index post consumption of 24 g freeze-dried dragon fruit.
Number of volunteers with treatment-related adverse events | Baseline & 12 weeks
  The number of volunteers with treatment-related adverse events will be assessed by questionnaires and interviews.

OTHER OUTCOMES:
Plasma and urine betalains and (poly)phenol metabolites | Baseline and 3 hours and 2 weeks post consumption
  Measured by liquid chromotography- mass spectrometry (LC/MS) post consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Rodriguez-Mateos, PhD, Principal Investigator — King's College London
Locations (1):
- King's College London, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheok A, Xu Y, Zhang Z, Caton PW, Rodriguez-Mateos A. Betalain-rich dragon fruit (pitaya) consumption improves vascular function in men and women: a double-blind, randomized controlled crossover trial. Am J Clin Nutr. 2022 May 1;115(5):1418-1431. doi: 10.1093/ajcn/nqab410. PMID 35265960